CLINICAL TRIAL: NCT00759291
Title: The Impact of Free Fatty Acid Reduction on Vascular Function in the Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua A. Beckman, MD, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2005P-001861
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Metabolic Syndrome
Keywords: free fatty acids; insulin-mediated; endothelium-dependent vasodilation; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acipimox (Active Comparator): Acipimox treatment QID for 7 days
  Interventions: Drug: acipimox
- Placebo (Placebo Comparator): Placebo treatment QID for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: acipimox — 250 mg tablet orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit
  Other Names: Olbetam
  Arms: Acipimox
Drug: Placebo — 1 tablet orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit
  Arms: Placebo

SUMMARY:
This study will test the hypothesis that reducing the release of free fatty acids (FFA) from fat cells will restore insulin-mediated, endothelium-dependent vasodilation in people with the metabolic syndrome.

DETAILED DESCRIPTION:
We hypothesize that acipimox, by decreasing plasma FFA concentrations, will augment endothelium-dependent vasodilation in conduit vessels and insulin-mediated vasodilation in forearm resistance arterioles in vivo, whole-body insulin sensitivity, and AKT (also known as Protein Kinase B) and endothelial nitric oxide synthase (eNOS) phosphorylation in skin biopsy specimens ex vivo, when compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults with metabolic syndrome, defined as the presence of 3 of 5 components of the syndrome as defined by the National Cholesterol Education Program including:

  * abdominal obesity
  * elevated fasting blood sugar (110 mg/dL< glucose < 126 mg/dL)
  * low HDL
  * elevated fasting blood triglycerides (> 150 mg/dL)
  * hypertension (BP > 140/90 mm HG)
* Normal cardiovascular examination

Exclusion Criteria:

* Diabetes mellitus
* Untreated hypercholesterolemia (LDL > 75th percentile for age)
* Cigarette smoking within 1 year
* Renal insufficiency (creatinine > 1.4 mg/dl)
* Blood dyscrasia
* Hepatic dysfunction (ALT > 2x normal)
* Evident coronary/peripheral atherosclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A. Beckman, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aday AW, Goldfine AB, Gregory JM, Beckman JA. Impact of Acipimox Therapy on Free Fatty Acid Efflux and Endothelial Function in the Metabolic Syndrome: A Randomized Trial. Obesity (Silver Spring). 2019 Nov;27(11):1812-1819. doi: 10.1002/oby.22602. Epub 2019 Oct 1. PMID 31571412
- [Derived] Sullivan AE, Courvan MCS, Ada AW, Wasserman DH, Niswender KD, Shardelow EM, Wells EK, Wells QS, Freiberg MS, Beckman JA. The Role of Serum Free Fatty Acids in Endothelium-Dependent Microvascular Function. Endocrinol Diabetes Metab. 2025 Mar;8(2):e70031. doi: 10.1002/edm2.70031. PMID 39888728

RESULTS

PARTICIPANT FLOW:
Groups:
- Acipimox First, Then Placebo: Acipimox treatment QID for 7 days, followed by a 4 week washout, and then Placebo treatment QID for 7 days.
  Acipimox: 250 mg tablet orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit.
  Placebo: 250 mg placebo tablets orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit.
- Placebo First, Then Acipimox: Placebo treatment QID for 7 days, followed by a four week washout, and then acipimox treatment for 7 day.
  Placebo: 250 mg placebo tablets orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit.
  Four week washout.
  Acipimox treatment QID for 7 days, followed by a 4 week washout, and then Placebo treatment QID for 7 days.
Period: First Treatment Period
Arm/Group | Acipimox First, Then Placebo | Placebo First, Then Acipimox
Started | 17 | 23
Completed | 17 | 23
Not Completed | 0 | 0
Period: Crossover
Arm/Group | Acipimox First, Then Placebo | Placebo First, Then Acipimox
Started | 17 (All subjects received acipicmox in the first period then received placebo in the second.) | 23 (All subjects who received placebo in the first period received acipimox in the second period.)
Completed | 17 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover trial in non diabetic subjects with and without the metabolic syndrome.
Groups:
- Acipimox First: Acipimox treatment QID for 7 days
  Acipimox: 250 mg tablet orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit
  then
  Placebo: 1 tablet orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit
- Placebo First: Placebo treatment QID for 7 days
  Placebo: 1 tablet orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit
  then
  Acipimox: 250 mg tablet orally every 6 hours for 7 days, with a dose at 7 am on the morning of the study visit
- Total: Total of all reporting groups
Arm/Group | Acipimox First | Placebo First | Total
Number analyzed (Participants) | 17 | 23 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 23 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (6) | 60 (11) | 56 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 10 | 15 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 23 | 40

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Vasodilation
Description: Brachial artery response to a 5 minute blood pressure cuff-applied ischemic period
Time Frame: After 7 days of each treatment.
Measure: Mean (Standard Deviation); unit: percentage of vasodilation
Groups:
- Metabolic Syndrome: Subjects with 3 or more criteria for metabolic syndrome.
- Control: Subjects without metabolic syndrome
Arm/Group | Metabolic Syndrome | Control
Number analyzed (Participants) | 18 | 17
percentage of vasodilation
  Placebo | 9.5 (6.5) | 10.8 (4.9)
  Acipimox | 10.5 (6) | 10.9 (6.2)

ADVERSE EVENTS:
Time Frame: 3 months
Description: It does not differ
Arm/Group | Acipimox | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2008-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT00759291/Prot_SAP_ICF_000.pdf